CLINICAL TRIAL: NCT02233647
Title: Safety and Tolerability of Cocaine During Phendimetrazine Maintenance
Brief Title: Phendimetrazine and Cocaine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BED (IN) 29
Record Dates: First submitted 2014-09-03; First posted 2014-09-08 (Estimated); Results first posted 2016-09-15 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Cocaine Use Disorder
Keywords: cocaine; phendimetrazine; pharmacotherapy
MeSH Terms: interventions — Cocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects will be maintained on oral placebo. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo
- Phendimetrazine Dose 1 (Experimental): Subjects will be maintained on the low phendimetrazine dose. Cocaine will be administered acutely during low dose phendimetrazine maintenance.
  Placebo will be administered acutely during low dose phendimetrazine maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo
- Phendimetrazine Dose 2 (Experimental): Subjects will be maintained on the intermediate phendimetrazine dose. Cocaine will be administered acutely during intermediate dose phendimetrazine maintenance.
  Placebo will be administered acutely during intermediate dose phendimetrazine maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo
- Phendimetrazine Dose 3 (Experimental): Subjects will be maintained on the high phendimetrazine dose. Cocaine will be administered acutely during high dose phendimetrazine maintenance.
  Placebo will be administered acutely during high dose phendimetrazine maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo

INTERVENTIONS:
Drug: Cocaine — The pharmacodynamic effects of cocaine will be determined during maintenance on placebo and phendimetrazine.
Drug: Placebo — The pharmacodynamic effects of placebo will be determined during maintenance on placebo and phendimetrazine.

SUMMARY:
This study will determine the safety and tolerability of phendimetrazine (Bontril®) as a pharmacotherapy for cocaine use disorder. A rigorous, inpatient human laboratory study will be conducted in which the subjective and physiological effects of cocaine are evaluated during maintenance on placebo and phendimetrazine.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine or phendimetrazine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven subjects were enrolled (i.e., signed consent), but only 10 subjects completed. Due to the within-subject nature of this study (i.e., missing data from the 11th subject cannot be analyzed with repeated-measures ANOVA), only data from the 10 subjects who completed the protocol were analyzed and reported.
Groups:
- Phendimetrazine Dose Escalation: Subjects were maintained on oral placebo, 70 mg phendimetrazine/day, 140 mg phendimetrazine/day and 210 mg phendimetrazine/day in ascending order.
  Intranasal cocaine (10, 20, 40 and 80 mg) was administered acutely after at least seven days of maintenance on each condition.
  Intransasal placebo cocaine was administered acutely after at least seven days of maintenance on each condition.
  Cocaine: The pharmacodynamic effects of cocaine were determined during maintenance on placebo and phendimetrazine.
  Placebo: The pharmacodynamic effects of placebo were determined during maintenance on placebo and phendimetrazine.
Period: Overall Study
Arm/Group | Phendimetrazine Dose Escalation
Started | 11
0 mg Cocaine With 0 mg Phendimetrazine | 11
10 mg Cocaine With 0 mg Phendimetrazine | 11
20 mg Cocaine With 0 mg Phendimetrazine | 10
40 mg Cocaine With 0 mg Phendimetrazine | 10
80 mg Cocaine With 0 mg Phendimetrazine | 10
0 mg Cocaine With 70 mg Phendimetrazine | 10
10 mg Cocaine With 70 mg Phendimetrazine | 10
20 mg Cocaine With 70 mg Phendimetrazine | 10
40 mg Cocaine With 70 mg Phendimetrazine | 10
80 mg Cocaine With 70 mg Phendimetrazine | 10
0 mg Cocaine With 140 mg Phendimetrazine | 10
10 mg Cocaine with140 mg Phendimetrazine | 10
20 mg Cocaine with140 mg Phendimetrazine | 10
40 mg Cocaine with140 mg Phendimetrazine | 10
80 mg Cocaine with140 mg Phendimetrazine | 10
0 mg Cocaine With 210 mg Phendimetrazine | 10
10 mg Cocaine with210 mg Phendimetrazine | 10
20 mg Cocaine with210 mg Phendimetrazine | 10
40 mg Cocaine with210 mg Phendimetrazine | 10
80 mg Cocaine with210 mg Phendimetrazine | 10
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: These are data for completing subjects only. Eleven subjects were enrolled (i.e., signed consent), but only data from completing subjects were included here and in the outcomes listed throughout this report.
Groups:
- Phendimetrazine Dose Escalation: Subjects were maintained on oral placebo, 70 mg phendimetrazine/day, 140 mg phendimetrazine/day and 210 mg phendimetrazine/day in ascending order.
  Cocaine was administered acutely after at least seven days of maintenance on each condition.
  Placebo cocaine was administered acutely after at least seven days of maintenance on each condition.
  Cocaine: The pharmacodynamic effects of cocaine were determined during maintenance on placebo and phendimetrazine.
  Placebo: The pharmacodynamic effects of placebo cocaine were determined during maintenance on placebo and phendimetrazine.
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Peak Systolic Pressure
Description: Systolic blood pressure was measured with an automated monitor. Higher values represent greater systolic pressure. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo maintenance conditions.
Time Frame: This measure was completed at 15 minute intervals after sampling each cocaine dose under both phendimetrazine and placebo maintenance conditions.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
mm Hg
  0 mg Cocaine with 0 mg Phendimetrazine | 115.4 (2.54)
  10 mg Cocaine with 0 mg Phendimetrazine | 121.3 (3.51)
  20 mg Cocaine with 0 mg Phendimetrazine | 123.4 (4.06)
  40 mg Cocaine with 0 mg Phendimetrazine | 122.1 (2.86)
  80 mg Cocaine with 0 mg Phendimetrazine | 135.4 (3.89)
  0 mg Cocaine with 70 mg Phendimetrazine | 120.0 (7.14)
  10 mg Cocaine with 70 mg Phendimetrazine | 119.7 (3.54)
  20 mg Cocaine with 70 mg Phendimetrazine | 119.9 (3.8)
  40 mg Cocaine with 70 mg Phendimetrazine | 125.4 (6.05)
  80 mg Cocaine with 70 mg Phendimetrazine | 130.3 (2.9)
  0 mg Cocaine with 140 mg Phendimetrazine | 117.9 (4.78)
  10 mg Cocaine with 140 mg Phendimetrazine | 121.7 (4.73)
  20 mg Cocaine with 140 mg Phendimetrazine | 122.1 (4.4)
  40 mg Cocaine with 140 mg Phendimetrazine | 121.5 (4.51)
  80 mg Cocaine with 140 mg Phendimetrazine | 131.9 (3.6)
  0 mg Cocaine with 210 mg Phendimetrazine | 119.2 (3.45)
  10 mg Cocaine with 210 mg Phendimetrazine | 119.7 (4.09)
  20 mg Cocaine with 210 mg Phendimetrazine | 119.8 (2.65)
  40 mg Cocaine with 210 mg Phendimetrazine | 119.3 (2.72)
  80 mg Cocaine with 210 mg Phendimetrazine | 130.9 (2.95)

2. Primary Outcome: Peak Diastolic Pressure
Description: Diastolic blood pressure was measured with an automated monitor. Higher values represent greater diastolic pressure. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo maintenance conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
mm Hg
  0 mg Cocaine with 0 mg Phendimetrazine | 75.6 (1.28)
  10 mg Cocaine with 0 mg Phendimetrazine | 75.2 (1.63)
  20 mg Cocaine with 0 mg Phendimetrazine | 78.4 (1.88)
  40 mg Cocaine with 0 mg Phendimetrazine | 78 (1.38)
  80 mg Cocaine with 0 mg Phendimetrazine | 80.8 (1.87)
  0 mg Cocaine with 70 mg Phendimetrazine | 77.2 (2.7)
  10 mg Cocaine with 70 mg Phendimetrazine | 76.7 (2.62)
  20 mg Cocaine with 70 mg Phendimetrazine | 75.6 (2.45)
  40 mg Cocaine with 70 mg Phendimetrazine | 75.6 (3.02)
  80 mg Cocaine with 70 mg Phendimetrazine | 83.2 (2.69)
  0 mg Cocaine with 140 mg Phendimetrazine | 74.3 (1.72)
  10 mg Cocaine with 140 mg Phendimetrazine | 76 (1.84)
  20 mg Cocaine with 140 mg Phendimetrazine | 78.1 (1.29)
  40 mg Cocaine with 140 mg Phendimetrazine | 77.7 (2.28)
  80 mg Cocaine with 140 mg Phendimetrazine | 83.6 (1.26)
  0 mg Cocaine with 210 mg Phendimetrazine | 76.6 (2.42)
  10 mg Cocaine with 210 mg Phendimetrazine | 77.9 (1.99)
  20 mg Cocaine with 210 mg Phendimetrazine | 80.7 (2.34)
  40 mg Cocaine with 210 mg Phendimetrazine | 78.6 (1.83)
  80 mg Cocaine with 210 mg Phendimetrazine | 84.8 (2.37)

3. Primary Outcome: Peak Heart Rate
Description: Heart rate was measured with an automated monitor. Higher values represent greater heart rate. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo maintenance conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Beats per Minute
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
Beats per Minute
  0 mg Cocaine with 0 mg Phendimetrazine | 75 (3.72)
  10 mg Cocaine with 0 mg Phendimetrazine | 72.7 (2.64)
  20 mg Cocaine with 0 mg Phendimetrazine | 77.4 (4.19)
  40 mg Cocaine with 0 mg Phendimetrazine | 79.2 (4.63)
  80 mg Cocaine with 0 mg Phendimetrazine | 87.8 (5.6)
  0 mg Cocaine with 70 mg Phendimetrazine | 76.6 (2.57)
  10 mg Cocaine with 70 mg Phendimetrazine | 75.3 (3.21)
  20 mg Cocaine with 70 mg Phendimetrazine | 77 (3.06)
  40 mg Cocaine with 70 mg Phendimetrazine | 81 (4.48)
  80 mg Cocaine with 70 mg Phendimetrazine | 83.8 (3.92)
  0 mg Cocaine with 140 mg Phendimetrazine | 82.1 (4.07)
  10 mg Cocaine with 140 mg Phendimetrazine | 81.1 (3.87)
  20 mg Cocaine with 140 mg Phendimetrazine | 83.4 (4.81)
  40 mg Cocaine with 140 mg Phendimetrazine | 83.5 (3.66)
  80 mg Cocaine with 140 mg Phendimetrazine | 84.8 (4.03)
  0 mg Cocaine with 210 mg Phendimetrazine | 84.9 (2.28)
  10 mg Cocaine with 210 mg Phendimetrazine | 77.5 (2.2)
  20 mg Cocaine with 210 mg Phendimetrazine | 85.3 (4.05)
  40 mg Cocaine with 210 mg Phendimetrazine | 82.8 (3.08)
  80 mg Cocaine with 210 mg Phendimetrazine | 88.9 (4.13)

4. Primary Outcome: Peak Temperature
Description: Oral temperature was measured with an automated monitor. Higher values represent greater temperature. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo maintenance conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Degrees Fahrenheit
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
Degrees Fahrenheit
  0 mg Cocaine with 0 mg Phendimetrazine | 98.09 (.13)
  10 mg Cocaine with 0 mg Phendimetrazine | 98.12 (.17)
  20 mg Cocaine with 0 mg Phendimetrazine | 98.24 (.12)
  40 mg Cocaine with 0 mg Phendimetrazine | 98.21 (.15)
  80 mg Cocaine with 0 mg Phendimetrazine | 98.04 (.29)
  0 mg Cocaine with 70 mg Phendimetrazine | 98.25 (.07)
  10 mg Cocaine with 70 mg Phendimetrazine | 98.28 (.08)
  20 mg Cocaine with 70 mg Phendimetrazine | 98.25 (.12)
  40 mg Cocaine with 70 mg Phendimetrazine | 98.24 (.22)
  80 mg Cocaine with 70 mg Phendimetrazine | 98.32 (.17)
  0 mg Cocaine with 140 mg Phendimetrazine | 98.19 (.04)
  10 mg Cocaine with 140 mg Phendimetrazine | 98.17 (.06)
  20 mg Cocaine with 140 mg Phendimetrazine | 98.25 (.05)
  40 mg Cocaine with 140 mg Phendimetrazine | 98.2 (.09)
  80 mg Cocaine with 140 mg Phendimetrazine | 98.3 (.04)
  0 mg Cocaine with 210 mg Phendimetrazine | 98.41 (.07)
  10 mg Cocaine with 210 mg Phendimetrazine | 98.17 (.06)
  20 mg Cocaine with 210 mg Phendimetrazine | 98.18 (.08)
  40 mg Cocaine with 210 mg Phendimetrazine | 98.24 (.07)
  80 mg Cocaine with 210 mg Phendimetrazine | 98.38 (.1)

5. Secondary Outcome: Peak Score on Sedative Subscale of the Adjective Rating Scale
Description: Subjects completed 16 items that loaded into the Sedative Subscale of the Adjective Rating Scale. The items were rated 0-4 on a Likert-type scale and the sum for the 16 "sedative" items was summed to yield the Sedative Subscale score. The maximum score for this scale was 64, the minimum was 0. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 2.3 (.68)
  10 mg Cocaine with 0 mg Phendimetrazine | 2.5 (.96)
  20 mg Cocaine with 0 mg Phendimetrazine | 2.5 (.99)
  40 mg Cocaine with 0 mg Phendimetrazine | 2.4 (.82)
  80 mg Cocaine with 0 mg Phendimetrazine | 4.4 (1.54)
  0 mg Cocaine with 70 mg Phendimetrazine | 1.9 (.59)
  10 mg Cocaine with 70 mg Phendimetrazine | 2.2 (1.03)
  20 mg Cocaine with 70 mg Phendimetrazine | 3.5 (1.65)
  40 mg Cocaine with 70 mg Phendimetrazine | 4.2 (2.27)
  80 mg Cocaine with 70 mg Phendimetrazine | 4.2 (2.06)
  0 mg Cocaine with 140 mg Phendimetrazine | 2.1 (1.22)
  10 mg Cocaine with 140 mg Phendimetrazine | 2.7 (1.56)
  20 mg Cocaine with 140 mg Phendimetrazine | 3.1 (1.62)
  40 mg Cocaine with 140 mg Phendimetrazine | 2.8 (1.52)
  80 mg Cocaine with 140 mg Phendimetrazine | 4.0 (2.19)
  0 mg Cocaine with 210 mg Phendimetrazine | 1.8 (.57)
  10 mg Cocaine with 210 mg Phendimetrazine | 2.6 (.9)
  20 mg Cocaine with 210 mg Phendimetrazine | 3.8 (1.4)
  40 mg Cocaine with 210 mg Phendimetrazine | 4.2 (1.68)
  80 mg Cocaine with 210 mg Phendimetrazine | 4.7 (2.26)

6. Secondary Outcome: Peak Score on Stimulant Subscale of the Adjective Rating Scale
Description: Subjects completed 16 items that loaded into the Stimulant Subscale of the Adjective Rating Scale. The items were rated 0-4 on a Likert-type scale and the sum for the 16 "stimulant" items was summed to yield the Stimulant Subscale score. The maximum score for this scale was 64, the minimum was 0. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 5.2 (1.05)
  10 mg Cocaine with 0 mg Phendimetrazine | 5.5 (1.33)
  20 mg Cocaine with 0 mg Phendimetrazine | 6.3 (1.52)
  40 mg Cocaine with 0 mg Phendimetrazine | 6.6 (1.64)
  80 mg Cocaine with 0 mg Phendimetrazine | 8.1 (1.47)
  0 mg Cocaine with 70 mg Phendimetrazine | 4.4 (.97)
  10 mg Cocaine with 70 mg Phendimetrazine | 5.2 (.92)
  20 mg Cocaine with 70 mg Phendimetrazine | 6.3 (1.17)
  40 mg Cocaine with 70 mg Phendimetrazine | 6.2 (.9)
  80 mg Cocaine with 70 mg Phendimetrazine | 7.3 (1.26)
  0 mg Cocaine with 140 mg Phendimetrazine | 3.7 (1.10)
  10 mg Cocaine with 140 mg Phendimetrazine | 5.3 (.91)
  20 mg Cocaine with 140 mg Phendimetrazine | 5.8 (1.18)
  40 mg Cocaine with 140 mg Phendimetrazine | 7.8 (1.54)
  80 mg Cocaine with 140 mg Phendimetrazine | 8.1 (1.43)
  0 mg Cocaine with 210 mg Phendimetrazine | 4.7 (1.08)
  10 mg Cocaine with 210 mg Phendimetrazine | 5.2 (1.14)
  20 mg Cocaine with 210 mg Phendimetrazine | 7.4 (1.38)
  40 mg Cocaine with 210 mg Phendimetrazine | 7.3 (1.35)
  80 mg Cocaine with 210 mg Phendimetrazine | 9 (1.23)

7. Secondary Outcome: Peak Ratings of "Active, Alert, Energetic" on the Visual Analog Scale
Description: Subjects rated their feelings of "Active, Alert, Energetic" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .6 (.5)
  10 mg Cocaine with 0 mg Phendimetrazine | 3.9 (1.91)
  20 mg Cocaine with 0 mg Phendimetrazine | 8.9 (3.89)
  40 mg Cocaine with 0 mg Phendimetrazine | 7.8 (4.99)
  80 mg Cocaine with 0 mg Phendimetrazine | 14 (6.23)
  0 mg Cocaine with 70 mg Phendimetrazine | 1.5 (1)
  10 mg Cocaine with 70 mg Phendimetrazine | 6 (2.28)
  20 mg Cocaine with 70 mg Phendimetrazine | 9 (3.87)
  40 mg Cocaine with 70 mg Phendimetrazine | 13.4 (3.91)
  80 mg Cocaine with 70 mg Phendimetrazine | 16 (4.17)
  0 mg Cocaine with 140 mg Phendimetrazine | .7 (.6)
  10 mg Cocaine with 140 mg Phendimetrazine | 4 (1.76)
  20 mg Cocaine with 140 mg Phendimetrazine | 11.4 (4.7)
  40 mg Cocaine with 140 mg Phendimetrazine | 14.8 (4.7)
  80 mg Cocaine with 140 mg Phendimetrazine | 18.9 (5.31)
  0 mg Cocaine with 210 mg Phendimetrazine | 1 (.89)
  10 mg Cocaine with 210 mg Phendimetrazine | 1.8 (.85)
  20 mg Cocaine with 210 mg Phendimetrazine | 10.1 (3.71)
  40 mg Cocaine with 210 mg Phendimetrazine | 11.1 (3.89)
  80 mg Cocaine with 210 mg Phendimetrazine | 17 (5.8)

8. Secondary Outcome: Peak Ratings of "Any Effect" on the Visual Analog Scale
Description: Subjects rated their feelings of "Any Effect" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1.5 (.83)
  10 mg Cocaine with 0 mg Phendimetrazine | 4.7 (1.57)
  20 mg Cocaine with 0 mg Phendimetrazine | 13.2 (4.93)
  40 mg Cocaine with 0 mg Phendimetrazine | 16.9 (4.32)
  80 mg Cocaine with 0 mg Phendimetrazine | 26 (6.53)
  0 mg Cocaine with 70 mg Phendimetrazine | .9 (.64)
  10 mg Cocaine with 70 mg Phendimetrazine | 7.7 (2.59)
  20 mg Cocaine with 70 mg Phendimetrazine | 13.5 (4.84)
  40 mg Cocaine with 70 mg Phendimetrazine | 21.2 (6.9)
  80 mg Cocaine with 70 mg Phendimetrazine | 27.3 (7.81)
  0 mg Cocaine with 140 mg Phendimetrazine | .5 (.5)
  10 mg Cocaine with 140 mg Phendimetrazine | 7 (1.99)
  20 mg Cocaine with 140 mg Phendimetrazine | 12.8 (3.59)
  40 mg Cocaine with 140 mg Phendimetrazine | 19 (4.96)
  80 mg Cocaine with 140 mg Phendimetrazine | 28.1 (4.86)
  0 mg Cocaine with 210 mg Phendimetrazine | 4.6 (2.74)
  10 mg Cocaine with 210 mg Phendimetrazine | 10.5 (3.37)
  20 mg Cocaine with 210 mg Phendimetrazine | 14.7 (4.33)
  40 mg Cocaine with 210 mg Phendimetrazine | 21.5 (4.25)
  80 mg Cocaine with 210 mg Phendimetrazine | 35.1 (7.54)

9. Secondary Outcome: Peak Ratings of "Bad Effect" on the Visual Analog Scale
Description: Subjects rated their feelings of "Bad Effect" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .6 (.4)
  10 mg Cocaine with 0 mg Phendimetrazine | 2.1 (1.3)
  20 mg Cocaine with 0 mg Phendimetrazine | 4.9 (3.52)
  40 mg Cocaine with 0 mg Phendimetrazine | 6.6 (4.04)
  80 mg Cocaine with 0 mg Phendimetrazine | 8.5 (4.74)
  0 mg Cocaine with 70 mg Phendimetrazine | 1.3 (.87)
  10 mg Cocaine with 70 mg Phendimetrazine | 2 (1.42)
  20 mg Cocaine with 70 mg Phendimetrazine | 5.6 (2.4)
  40 mg Cocaine with 70 mg Phendimetrazine | 4.9 (2.70)
  80 mg Cocaine with 70 mg Phendimetrazine | 5.6 (3.73)
  0 mg Cocaine with 140 mg Phendimetrazine | .7 (.7)
  10 mg Cocaine with 140 mg Phendimetrazine | 1.9 (1.33)
  20 mg Cocaine with 140 mg Phendimetrazine | 5.7 (3.14)
  40 mg Cocaine with 140 mg Phendimetrazine | 3.7 (2.63)
  80 mg Cocaine with 140 mg Phendimetrazine | 11.4 (5.39)
  0 mg Cocaine with 210 mg Phendimetrazine | 9.2 (7.77)
  10 mg Cocaine with 210 mg Phendimetrazine | 2.4 (1.52)
  20 mg Cocaine with 210 mg Phendimetrazine | 3.9 (2.17)
  40 mg Cocaine with 210 mg Phendimetrazine | 8.1 (4.45)
  80 mg Cocaine with 210 mg Phendimetrazine | 10.2 (7.23)

10. Secondary Outcome: Peak Ratings of "Euphoric" on the Visual Analog Scale
Description: Subjects rated their feelings of "Euphoric" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1 (.89)
  10 mg Cocaine with 0 mg Phendimetrazine | 1.8 (.87)
  20 mg Cocaine with 0 mg Phendimetrazine | 3.1 (1.87)
  40 mg Cocaine with 0 mg Phendimetrazine | 1.2 (.81)
  80 mg Cocaine with 0 mg Phendimetrazine | 1.9 (1.32)
  0 mg Cocaine with 70 mg Phendimetrazine | 1 (.6)
  10 mg Cocaine with 70 mg Phendimetrazine | 1 (.52)
  20 mg Cocaine with 70 mg Phendimetrazine | 3.2 (1.52)
  40 mg Cocaine with 70 mg Phendimetrazine | 1.2 (.63)
  80 mg Cocaine with 70 mg Phendimetrazine | 2 (1)
  0 mg Cocaine with 140 mg Phendimetrazine | .9 (.64)
  10 mg Cocaine with 140 mg Phendimetrazine | 2 (1.16)
  20 mg Cocaine with 140 mg Phendimetrazine | 1.3 (.7)
  40 mg Cocaine with 140 mg Phendimetrazine | 1 (.54)
  80 mg Cocaine with 140 mg Phendimetrazine | 1.3 (.7)
  0 mg Cocaine with 210 mg Phendimetrazine | .9 (.48)
  10 mg Cocaine with 210 mg Phendimetrazine | .4 (.4)
  20 mg Cocaine with 210 mg Phendimetrazine | 1 (.68)
  40 mg Cocaine with 210 mg Phendimetrazine | .8 (.47)
  80 mg Cocaine with 210 mg Phendimetrazine | 1.7 (.82)

11. Secondary Outcome: Peak Ratings of "Good Effect" on the Visual Analog Scale
Description: Subjects rated their feelings of "Good Effect" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1.2 (.73)
  10 mg Cocaine with 0 mg Phendimetrazine | 7.1 (2.74)
  20 mg Cocaine with 0 mg Phendimetrazine | 12.4 (4.61)
  40 mg Cocaine with 0 mg Phendimetrazine | 12.3 (5.27)
  80 mg Cocaine with 0 mg Phendimetrazine | 19.8 (7.01)
  0 mg Cocaine with 70 mg Phendimetrazine | 1.3 (.94)
  10 mg Cocaine with 70 mg Phendimetrazine | 7.1 (2.48)
  20 mg Cocaine with 70 mg Phendimetrazine | 11.7 (3.77)
  40 mg Cocaine with 70 mg Phendimetrazine | 15.3 (5.14)
  80 mg Cocaine with 70 mg Phendimetrazine | 21.3 (5.57)
  0 mg Cocaine with 140 mg Phendimetrazine | 2.1 (1.13)
  10 mg Cocaine with 140 mg Phendimetrazine | 8.1 (2.67)
  20 mg Cocaine with 140 mg Phendimetrazine | 7.9 (3.9)
  40 mg Cocaine with 140 mg Phendimetrazine | 15.4 (5.39)
  80 mg Cocaine with 140 mg Phendimetrazine | 27.8 (6.5)
  0 mg Cocaine with 210 mg Phendimetrazine | 9.2 (7.77)
  10 mg Cocaine with 210 mg Phendimetrazine | 12 (4.51)
  20 mg Cocaine with 210 mg Phendimetrazine | 16.7 (6.33)
  40 mg Cocaine with 210 mg Phendimetrazine | 17.1 (4.33)
  80 mg Cocaine with 210 mg Phendimetrazine | 27.2 (7.56)

12. Secondary Outcome: Peak Ratings of "High" on the Visual Analog Scale
Description: Subjects rated their feelings of "High" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1.4 (.69)
  10 mg Cocaine with 0 mg Phendimetrazine | 6 (2.29)
  20 mg Cocaine with 0 mg Phendimetrazine | 14.1 (4.9)
  40 mg Cocaine with 0 mg Phendimetrazine | 11.9 (4.81)
  80 mg Cocaine with 0 mg Phendimetrazine | 23.4 (6.42)
  0 mg Cocaine with 70 mg Phendimetrazine | 1.1 (.6)
  10 mg Cocaine with 70 mg Phendimetrazine | 3.6 (1.18)
  20 mg Cocaine with 70 mg Phendimetrazine | 10.8 (4.14)
  40 mg Cocaine with 70 mg Phendimetrazine | 13.3 (5.55)
  80 mg Cocaine with 70 mg Phendimetrazine | 18.6 (6.52)
  0 mg Cocaine with 140 mg Phendimetrazine | .6 (.5)
  10 mg Cocaine with 140 mg Phendimetrazine | 6.3 (2.96)
  20 mg Cocaine with 140 mg Phendimetrazine | 9.1 (4.39)
  40 mg Cocaine with 140 mg Phendimetrazine | 15.8 (5.96)
  80 mg Cocaine with 140 mg Phendimetrazine | 24.2 (6.77)
  0 mg Cocaine with 210 mg Phendimetrazine | .8 (.59)
  10 mg Cocaine with 210 mg Phendimetrazine | 8.3 (4.14)
  20 mg Cocaine with 210 mg Phendimetrazine | 15.3 (6.35)
  40 mg Cocaine with 210 mg Phendimetrazine | 12.1 (3.14)
  80 mg Cocaine with 210 mg Phendimetrazine | 22.6 (7.05)

13. Secondary Outcome: Peak Ratings of "Irregular/Racing Heartbeat" on the Visual Analog Scale
Description: Subjects rated their feelings of "Irregular/Racing Heartbeat" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .8 (.51)
  10 mg Cocaine with 0 mg Phendimetrazine | 2.8 (1.19)
  20 mg Cocaine with 0 mg Phendimetrazine | 10.8 (4.07)
  40 mg Cocaine with 0 mg Phendimetrazine | 9.2 (5)
  80 mg Cocaine with 0 mg Phendimetrazine | 14.6 (7)
  0 mg Cocaine with 70 mg Phendimetrazine | .4 (.4)
  10 mg Cocaine with 70 mg Phendimetrazine | 1.6 (.6)
  20 mg Cocaine with 70 mg Phendimetrazine | 6.9 (3.7)
  40 mg Cocaine with 70 mg Phendimetrazine | 2.4 (1.3)
  80 mg Cocaine with 70 mg Phendimetrazine | 6 (2.9)
  0 mg Cocaine with 140 mg Phendimetrazine | .6 (.4)
  10 mg Cocaine with 140 mg Phendimetrazine | .8 (.55)
  20 mg Cocaine with 140 mg Phendimetrazine | 3.6 (2.56)
  40 mg Cocaine with 140 mg Phendimetrazine | 5.10 (2.15)
  80 mg Cocaine with 140 mg Phendimetrazine | 8.2 (4.17)
  0 mg Cocaine with 210 mg Phendimetrazine | 2.3 (1.21)
  10 mg Cocaine with 210 mg Phendimetrazine | .6 (.5)
  20 mg Cocaine with 210 mg Phendimetrazine | 4 (3.36)
  40 mg Cocaine with 210 mg Phendimetrazine | 5.5 (3.48)
  80 mg Cocaine with 210 mg Phendimetrazine | 9.8 (4.85)

14. Secondary Outcome: Peak Ratings of "Like Drug" on the Visual Analog Scale
Description: Subjects rated their feelings of "Like Drug" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1 (.54)
  10 mg Cocaine with 0 mg Phendimetrazine | 6.4 (2.01)
  20 mg Cocaine with 0 mg Phendimetrazine | 12.9 (4.58)
  40 mg Cocaine with 0 mg Phendimetrazine | 14 (5.82)
  80 mg Cocaine with 0 mg Phendimetrazine | 23.2 (8.32)
  0 mg Cocaine with 70 mg Phendimetrazine | .5 (.5)
  10 mg Cocaine with 70 mg Phendimetrazine | 4.1 (1.49)
  20 mg Cocaine with 70 mg Phendimetrazine | 10.7 (3.52)
  40 mg Cocaine with 70 mg Phendimetrazine | 17.9 (5.13)
  80 mg Cocaine with 70 mg Phendimetrazine | 25 (6.93)
  0 mg Cocaine with 140 mg Phendimetrazine | 1.2 (.8)
  10 mg Cocaine with 140 mg Phendimetrazine | 9.8 (3.16)
  20 mg Cocaine with 140 mg Phendimetrazine | 9.9 (3.93)
  40 mg Cocaine with 140 mg Phendimetrazine | 18 (6.01)
  80 mg Cocaine with 140 mg Phendimetrazine | 26.2 (6.32)
  0 mg Cocaine with 210 mg Phendimetrazine | 2.2 (1.44)
  10 mg Cocaine with 210 mg Phendimetrazine | 7.5 (2.66)
  20 mg Cocaine with 210 mg Phendimetrazine | 13.1 (4.72)
  40 mg Cocaine with 210 mg Phendimetrazine | 25.5 (9.3)
  80 mg Cocaine with 210 mg Phendimetrazine | 26.5 (8.32)

15. Secondary Outcome: Peak Ratings of "Nauseated/Queasy/Sick to Stomach" on the Visual Analog Scale
Description: Subjects rated their feelings of "Nauseated/Queasy/Sick to Stomach" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1.4 (.69)
  10 mg Cocaine with 0 mg Phendimetrazine | 3.3 (1.54)
  20 mg Cocaine with 0 mg Phendimetrazine | 3.1 (1.29)
  40 mg Cocaine with 0 mg Phendimetrazine | 7.8 (2.59)
  80 mg Cocaine with 0 mg Phendimetrazine | 14 (5.79)
  0 mg Cocaine with 70 mg Phendimetrazine | .6 (.43)
  10 mg Cocaine with 70 mg Phendimetrazine | 4.3 (2.32)
  20 mg Cocaine with 70 mg Phendimetrazine | 4.3 (2.17)
  40 mg Cocaine with 70 mg Phendimetrazine | 5.3 (4.22)
  80 mg Cocaine with 70 mg Phendimetrazine | 10.5 (5.45)
  0 mg Cocaine with 140 mg Phendimetrazine | .6 (.5)
  10 mg Cocaine with 140 mg Phendimetrazine | 4.1 (2.77)
  20 mg Cocaine with 140 mg Phendimetrazine | 2.9 (1.96)
  40 mg Cocaine with 140 mg Phendimetrazine | 6.9 (3.59)
  80 mg Cocaine with 140 mg Phendimetrazine | 10.7 (5.7)
  0 mg Cocaine with 210 mg Phendimetrazine | 5.2 (4.14)
  10 mg Cocaine with 210 mg Phendimetrazine | 1.7 (1.25)
  20 mg Cocaine with 210 mg Phendimetrazine | 4.8 (2.83)
  40 mg Cocaine with 210 mg Phendimetrazine | 4.3 (2.54)
  80 mg Cocaine with 210 mg Phendimetrazine | 2.9 (1.89)

16. Secondary Outcome: Peak Ratings of "Nervous/Anxious" on the Visual Analog Scale
Description: Subjects rated their feelings of "Nervous/Anxious" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .7 (.47)
  10 mg Cocaine with 0 mg Phendimetrazine | 2.3 (1.12)
  20 mg Cocaine with 0 mg Phendimetrazine | 3.7 (2.27)
  40 mg Cocaine with 0 mg Phendimetrazine | 4.1 (2.61)
  80 mg Cocaine with 0 mg Phendimetrazine | 9.4 (6)
  0 mg Cocaine with 70 mg Phendimetrazine | .6 (.43)
  10 mg Cocaine with 70 mg Phendimetrazine | .9 (.53)
  20 mg Cocaine with 70 mg Phendimetrazine | 2 (1.14)
  40 mg Cocaine with 70 mg Phendimetrazine | 5.4 (2.50)
  80 mg Cocaine with 70 mg Phendimetrazine | 7.7 (4.46)
  0 mg Cocaine with 140 mg Phendimetrazine | .5 (.4)
  10 mg Cocaine with 140 mg Phendimetrazine | 1.7 (.75)
  20 mg Cocaine with 140 mg Phendimetrazine | 2.5 (1.24)
  40 mg Cocaine with 140 mg Phendimetrazine | 6.7 (2.96)
  80 mg Cocaine with 140 mg Phendimetrazine | 10.5 (4.22)
  0 mg Cocaine with 210 mg Phendimetrazine | .8 (.55)
  10 mg Cocaine with 210 mg Phendimetrazine | .5 (.4)
  20 mg Cocaine with 210 mg Phendimetrazine | 3.7 (2.13)
  40 mg Cocaine with 210 mg Phendimetrazine | 4.4 (2.28)
  80 mg Cocaine with 210 mg Phendimetrazine | 10.1 (6.52)

17. Secondary Outcome: Peak Ratings of "Willing to Pay For" on the Visual Analog Scale
Description: Subjects rated their feelings of "Willing to Pay For" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .9 (.9)
  10 mg Cocaine with 0 mg Phendimetrazine | 4.4 (2.49)
  20 mg Cocaine with 0 mg Phendimetrazine | 8.2 (3.53)
  40 mg Cocaine with 0 mg Phendimetrazine | 11.2 (4.59)
  80 mg Cocaine with 0 mg Phendimetrazine | 20.2 (7.01)
  0 mg Cocaine with 70 mg Phendimetrazine | 1.1 (.72)
  10 mg Cocaine with 70 mg Phendimetrazine | 1.4 (.86)
  20 mg Cocaine with 70 mg Phendimetrazine | 6.4 (2.9)
  40 mg Cocaine with 70 mg Phendimetrazine | 14.1 (4.62)
  80 mg Cocaine with 70 mg Phendimetrazine | 19.3 (5.63)
  0 mg Cocaine with 140 mg Phendimetrazine | .8 (.42)
  10 mg Cocaine with 140 mg Phendimetrazine | 3.2 (2.15)
  20 mg Cocaine with 140 mg Phendimetrazine | 7.9 (3.82)
  40 mg Cocaine with 140 mg Phendimetrazine | 18.3 (6.58)
  80 mg Cocaine with 140 mg Phendimetrazine | 23 (5.77)
  0 mg Cocaine with 210 mg Phendimetrazine | 1.7 (1.32)
  10 mg Cocaine with 210 mg Phendimetrazine | 6 (2.65)
  20 mg Cocaine with 210 mg Phendimetrazine | 8.9 (4.39)
  40 mg Cocaine with 210 mg Phendimetrazine | 12.3 (3.77)
  80 mg Cocaine with 210 mg Phendimetrazine | 23.1 (9.27)

18. Secondary Outcome: Peak Ratings of "Performance Impaired" on the Visual Analog Scale
Description: Subjects rated their feelings of "Performance Impaired" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .8 (.7)
  10 mg Cocaine with 0 mg Phendimetrazine | .7 (.47)
  20 mg Cocaine with 0 mg Phendimetrazine | 1.9 (.98)
  40 mg Cocaine with 0 mg Phendimetrazine | 3.3 (1.24)
  80 mg Cocaine with 0 mg Phendimetrazine | 3.4 (1.31)
  0 mg Cocaine with 70 mg Phendimetrazine | 1 (.68)
  10 mg Cocaine with 70 mg Phendimetrazine | 2.2 (1.12)
  20 mg Cocaine with 70 mg Phendimetrazine | .8 (.55)
  40 mg Cocaine with 70 mg Phendimetrazine | .7 (.6)
  80 mg Cocaine with 70 mg Phendimetrazine | 4.9 (2.82)
  0 mg Cocaine with 140 mg Phendimetrazine | .8 (.42)
  10 mg Cocaine with 140 mg Phendimetrazine | .7 (.47)
  20 mg Cocaine with 140 mg Phendimetrazine | 4.5 (3.56)
  40 mg Cocaine with 140 mg Phendimetrazine | 2.1 (1)
  80 mg Cocaine with 140 mg Phendimetrazine | 3.7 (1.78)
  0 mg Cocaine with 210 mg Phendimetrazine | .8 (.55)
  10 mg Cocaine with 210 mg Phendimetrazine | .3 (.3)
  20 mg Cocaine with 210 mg Phendimetrazine | 7.6 (5.07)
  40 mg Cocaine with 210 mg Phendimetrazine | 4.4 (3.65)
  80 mg Cocaine with 210 mg Phendimetrazine | 7.6 (5.24)

19. Secondary Outcome: Peak Ratings of "Performance Improved" on the Visual Analog Scale
Description: Subjects rated their feelings of "Performance Improved" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .7 (.6)
  10 mg Cocaine with 0 mg Phendimetrazine | .7 (.42)
  20 mg Cocaine with 0 mg Phendimetrazine | 1.4 (.72)
  40 mg Cocaine with 0 mg Phendimetrazine | 1.4 (.6)
  80 mg Cocaine with 0 mg Phendimetrazine | 6.6 (4.49)
  0 mg Cocaine with 70 mg Phendimetrazine | .7 (.6)
  10 mg Cocaine with 70 mg Phendimetrazine | .6 (.5)
  20 mg Cocaine with 70 mg Phendimetrazine | 1.9 (.91)
  40 mg Cocaine with 70 mg Phendimetrazine | 4.8 (3.31)
  80 mg Cocaine with 70 mg Phendimetrazine | 2.4 (1.15)
  0 mg Cocaine with 140 mg Phendimetrazine | .9 (.6)
  10 mg Cocaine with 140 mg Phendimetrazine | .9 (.6)
  20 mg Cocaine with 140 mg Phendimetrazine | .8 (.61)
  40 mg Cocaine with 140 mg Phendimetrazine | 3.6 (2.84)
  80 mg Cocaine with 140 mg Phendimetrazine | 5.1 (3.58)
  0 mg Cocaine with 210 mg Phendimetrazine | 1.9 (1.29)
  10 mg Cocaine with 210 mg Phendimetrazine | .5 (.4)
  20 mg Cocaine with 210 mg Phendimetrazine | 1.6 (1.06)
  40 mg Cocaine with 210 mg Phendimetrazine | 3.9 (2.9)
  80 mg Cocaine with 210 mg Phendimetrazine | 2.6 (1.65)

20. Secondary Outcome: Peak Ratings of "Restless" on the Visual Analog Scale
Description: Subjects rated their feelings of "Restless" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .5 (.4)
  10 mg Cocaine with 0 mg Phendimetrazine | 1.9 (1.08)
  20 mg Cocaine with 0 mg Phendimetrazine | .7 (.6)
  40 mg Cocaine with 0 mg Phendimetrazine | 1.8 (1.01)
  80 mg Cocaine with 0 mg Phendimetrazine | 2.3 (1.32)
  0 mg Cocaine with 70 mg Phendimetrazine | .5 (.5)
  10 mg Cocaine with 70 mg Phendimetrazine | .9 (.53)
  20 mg Cocaine with 70 mg Phendimetrazine | .7 (.47)
  40 mg Cocaine with 70 mg Phendimetrazine | 1.1 (.64)
  80 mg Cocaine with 70 mg Phendimetrazine | 1 (.54)
  0 mg Cocaine with 140 mg Phendimetrazine | 1 (.68)
  10 mg Cocaine with 140 mg Phendimetrazine | 1.8 (.9)
  20 mg Cocaine with 140 mg Phendimetrazine | 2.3 (1.67)
  40 mg Cocaine with 140 mg Phendimetrazine | 4.1 (1.96)
  80 mg Cocaine with 140 mg Phendimetrazine | 4 (2.04)
  0 mg Cocaine with 210 mg Phendimetrazine | 1.6 (.99)
  10 mg Cocaine with 210 mg Phendimetrazine | 2.7 (2.28)
  20 mg Cocaine with 210 mg Phendimetrazine | 2.0 (1.61)
  40 mg Cocaine with 210 mg Phendimetrazine | 3.6 (1.59)
  80 mg Cocaine with 210 mg Phendimetrazine | 6.9 (5.38)

21. Secondary Outcome: Peak Ratings of "Rush" on the Visual Analog Scale
Description: Subjects rated their feelings of "Rush" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | .5 (.5)
  10 mg Cocaine with 0 mg Phendimetrazine | 4.4 (2.4)
  20 mg Cocaine with 0 mg Phendimetrazine | 11.9 (4.53)
  40 mg Cocaine with 0 mg Phendimetrazine | 11.4 (5.93)
  80 mg Cocaine with 0 mg Phendimetrazine | 17.4 (7.06)
  0 mg Cocaine with 70 mg Phendimetrazine | .9 (.6)
  10 mg Cocaine with 70 mg Phendimetrazine | 3.4 (1.5)
  20 mg Cocaine with 70 mg Phendimetrazine | 8 (3.73)
  40 mg Cocaine with 70 mg Phendimetrazine | 11.1 (4.32)
  80 mg Cocaine with 70 mg Phendimetrazine | 20 (7.11)
  0 mg Cocaine with 140 mg Phendimetrazine | 1 (.67)
  10 mg Cocaine with 140 mg Phendimetrazine | 5.67 (2.12)
  20 mg Cocaine with 140 mg Phendimetrazine | 9.2 (3.44)
  40 mg Cocaine with 140 mg Phendimetrazine | 16.3 (5.95)
  80 mg Cocaine with 140 mg Phendimetrazine | 21.8 (6.03)
  0 mg Cocaine with 210 mg Phendimetrazine | 1.4 (.86)
  10 mg Cocaine with 210 mg Phendimetrazine | 7.3 (2.49)
  20 mg Cocaine with 210 mg Phendimetrazine | 10.3 (3.62)
  40 mg Cocaine with 210 mg Phendimetrazine | 13.2 (4.55)
  80 mg Cocaine with 210 mg Phendimetrazine | 16.9 (5.58)

22. Secondary Outcome: Peak Ratings of "Shaky/Jittery" on the Visual Analog Scale
Description: Subjects rated their feelings of "Shaky/Jittery" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1.7 (.88)
  10 mg Cocaine with 0 mg Phendimetrazine | 1.8 (.88)
  20 mg Cocaine with 0 mg Phendimetrazine | 6.1 (3.14)
  40 mg Cocaine with 0 mg Phendimetrazine | 6 (3.78)
  80 mg Cocaine with 0 mg Phendimetrazine | 11.9 (7.28)
  0 mg Cocaine with 70 mg Phendimetrazine | .4 (.4)
  10 mg Cocaine with 70 mg Phendimetrazine | .5 (.5)
  20 mg Cocaine with 70 mg Phendimetrazine | 1.8 (1.05)
  40 mg Cocaine with 70 mg Phendimetrazine | 2.4 (1.61)
  80 mg Cocaine with 70 mg Phendimetrazine | 6.5 (3.39)
  0 mg Cocaine with 140 mg Phendimetrazine | 1.4 (.79)
  10 mg Cocaine with 140 mg Phendimetrazine | .9 (.6)
  20 mg Cocaine with 140 mg Phendimetrazine | 3.8 (1.7)
  40 mg Cocaine with 140 mg Phendimetrazine | 3.9 (2.3)
  80 mg Cocaine with 140 mg Phendimetrazine | 12.8 (5.33)
  0 mg Cocaine with 210 mg Phendimetrazine | .3 (.3)
  10 mg Cocaine with 210 mg Phendimetrazine | .8 (.55)
  20 mg Cocaine with 210 mg Phendimetrazine | 1.9 (1.04)
  40 mg Cocaine with 210 mg Phendimetrazine | 6.6 (2.92)
  80 mg Cocaine with 210 mg Phendimetrazine | 9 (5.58)

23. Secondary Outcome: Peak Ratings of "Sluggish/Fatigued/Lazy" on the Visual Analog Scale
Description: Subjects rated their feelings of "Sluggish/Fatigued/Lazy" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1.7 (.9)
  10 mg Cocaine with 0 mg Phendimetrazine | 1.8 (1.09)
  20 mg Cocaine with 0 mg Phendimetrazine | 1.09 (1)
  40 mg Cocaine with 0 mg Phendimetrazine | 3.3 (1.81)
  80 mg Cocaine with 0 mg Phendimetrazine | 8.5 (5.85)
  0 mg Cocaine with 70 mg Phendimetrazine | .6 (.43)
  10 mg Cocaine with 70 mg Phendimetrazine | 3.0 (1.96)
  20 mg Cocaine with 70 mg Phendimetrazine | 3.3 (2.47)
  40 mg Cocaine with 70 mg Phendimetrazine | 5.3 (3.53)
  80 mg Cocaine with 70 mg Phendimetrazine | 6 (3.53)
  0 mg Cocaine with 140 mg Phendimetrazine | .7 (.4)
  10 mg Cocaine with 140 mg Phendimetrazine | 4.8 (2.27)
  20 mg Cocaine with 140 mg Phendimetrazine | 4.6 (2.47)
  40 mg Cocaine with 140 mg Phendimetrazine | 5.3 (2.94)
  80 mg Cocaine with 140 mg Phendimetrazine | 10.9 (5.49)
  0 mg Cocaine with 210 mg Phendimetrazine | 7 (5.82)
  10 mg Cocaine with 210 mg Phendimetrazine | 5.5 (2.67)
  20 mg Cocaine with 210 mg Phendimetrazine | 4.8 (2.64)
  40 mg Cocaine with 210 mg Phendimetrazine | 4.2 (2.63)
  80 mg Cocaine with 210 mg Phendimetrazine | 8.8 (7.16)

24. Secondary Outcome: Peak Ratings of "Stimulated" on the Visual Analog Scale
Description: Subjects rated their feelings of "Stimulated" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1.8 (.8)
  10 mg Cocaine with 0 mg Phendimetrazine | 2 (.93)
  20 mg Cocaine with 0 mg Phendimetrazine | 5.6 (2.9)
  40 mg Cocaine with 0 mg Phendimetrazine | 5.1 (2.56)
  80 mg Cocaine with 0 mg Phendimetrazine | 10.8 (4.92)
  0 mg Cocaine with 70 mg Phendimetrazine | .8 (.53)
  10 mg Cocaine with 70 mg Phendimetrazine | 3.7 (1.55)
  20 mg Cocaine with 70 mg Phendimetrazine | 4.9 (2.61)
  40 mg Cocaine with 70 mg Phendimetrazine | 8.9 (4.42)
  80 mg Cocaine with 70 mg Phendimetrazine | 12.4 (4.53)
  0 mg Cocaine with 140 mg Phendimetrazine | 1.6 (.82)
  10 mg Cocaine with 140 mg Phendimetrazine | 2.9 (1.28)
  20 mg Cocaine with 140 mg Phendimetrazine | 5.5 (3.59)
  40 mg Cocaine with 140 mg Phendimetrazine | 11.6 (5.36)
  80 mg Cocaine with 140 mg Phendimetrazine | 10.9 (5.12)
  0 mg Cocaine with 210 mg Phendimetrazine | 2.2 (1.14)
  10 mg Cocaine with 210 mg Phendimetrazine | 2.4 (1.56)
  20 mg Cocaine with 210 mg Phendimetrazine | 4.8 (2.45)
  40 mg Cocaine with 210 mg Phendimetrazine | 9.1 (3.52)
  80 mg Cocaine with 210 mg Phendimetrazine | 14.7 (6.91)

25. Secondary Outcome: Peak Ratings of "Willing to Take Again" on the Visual Analog Scale
Description: Subjects rated their feelings of "Willing to Take Again" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1.1 (.66)
  10 mg Cocaine with 0 mg Phendimetrazine | 9.8 (5.13)
  20 mg Cocaine with 0 mg Phendimetrazine | 14.1 (5.44)
  40 mg Cocaine with 0 mg Phendimetrazine | 16.5 (7.26)
  80 mg Cocaine with 0 mg Phendimetrazine | 22.9 (8.82)
  0 mg Cocaine with 70 mg Phendimetrazine | 1.5 (.89)
  10 mg Cocaine with 70 mg Phendimetrazine | 3.5 (.96)
  20 mg Cocaine with 70 mg Phendimetrazine | 13 (3.86)
  40 mg Cocaine with 70 mg Phendimetrazine | 20.7 (5.96)
  80 mg Cocaine with 70 mg Phendimetrazine | 26.7 (7.53)
  0 mg Cocaine with 140 mg Phendimetrazine | 1 (.63)
  10 mg Cocaine with 140 mg Phendimetrazine | 8.8 (4.12)
  20 mg Cocaine with 140 mg Phendimetrazine | 11.1 (4.8)
  40 mg Cocaine with 140 mg Phendimetrazine | 19.4 (5.81)
  80 mg Cocaine with 140 mg Phendimetrazine | 25.8 (5.2)
  0 mg Cocaine with 210 mg Phendimetrazine | 2 (1.32)
  10 mg Cocaine with 210 mg Phendimetrazine | 11.2 (5.20)
  20 mg Cocaine with 210 mg Phendimetrazine | 11.6 (4.69)
  40 mg Cocaine with 210 mg Phendimetrazine | 17.9 (5.15)
  80 mg Cocaine with 210 mg Phendimetrazine | 30 (8.78)

26. Secondary Outcome: Peak Ratings of "Talkative/Friendly" on the Visual Analog Scale
Description: Subjects rated their feelings of "Talkative/Friendly" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both phendimetrazine and placebo conditions.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phendimetrazine Dose Escalation
Number analyzed (Participants) | 10
units on a scale
  0 mg Cocaine with 0 mg Phendimetrazine | 1 (.6)
  10 mg Cocaine with 0 mg Phendimetrazine | 2.7 (1.28)
  20 mg Cocaine with 0 mg Phendimetrazine | 3.9 (2.96)
  40 mg Cocaine with 0 mg Phendimetrazine | 3.5 (2.4)
  80 mg Cocaine with 0 mg Phendimetrazine | 4.3 (2.82)
  0 mg Cocaine with 70 mg Phendimetrazine | .6 (.6)
  10 mg Cocaine with 70 mg Phendimetrazine | 2.7 (1.21)
  20 mg Cocaine with 70 mg Phendimetrazine | 5.4 (2.63)
  40 mg Cocaine with 70 mg Phendimetrazine | 7.3 (3.09)
  80 mg Cocaine with 70 mg Phendimetrazine | 8 (3.87)
  0 mg Cocaine with 140 mg Phendimetrazine | 1 (.68)
  10 mg Cocaine with 140 mg Phendimetrazine | 1.2 (.81)
  20 mg Cocaine with 140 mg Phendimetrazine | 1.9 (1.04)
  40 mg Cocaine with 140 mg Phendimetrazine | 3.2 (1.65)
  80 mg Cocaine with 140 mg Phendimetrazine | 7.2 (2.74)
  0 mg Cocaine with 210 mg Phendimetrazine | .7 (.47)
  10 mg Cocaine with 210 mg Phendimetrazine | .5 (.34)
  20 mg Cocaine with 210 mg Phendimetrazine | 1.9 (.92)
  40 mg Cocaine with 210 mg Phendimetrazine | 1.7 (1.11)
  80 mg Cocaine with 210 mg Phendimetrazine | 3.4 (1.43)

ADVERSE EVENTS:
Arm/Group | Phendimetrazine Dose Escalation
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phendimetrazine Dose Escalation (N=11)
Persistent Tachycardia (Cardiac disorders) | 1 (1) — One subject experienced persistent tachycardia after receiving 10 mg cocaine during placebo maintenance and was discharged from the protocol after the event resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No